CLINICAL TRIAL: NCT05010070
Title: The University of Michigan Wellness Education for Liver Health Study
Brief Title: The University of Michigan Wellness for Liver Health Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00154361
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: nutrition
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diet and lifestyle program (Experimental): Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep. They will also be taught about positive affect skills (such as gratitude, positive reappraisal, and personal strengths) and mindful eating.
  Interventions: Behavioral: diet and lifestyle program

INTERVENTIONS:
Behavioral: diet and lifestyle program — See description of main arm.

SUMMARY:
The goal of this proposal is to pilot test our existing very-low carbohydrate diet intervention, adapted for adults with Non-alcoholic Fatty Liver Disease (NAFLD).

DETAILED DESCRIPTION:
As there are no medications that effectively treat nonalcoholic fatty liver disease (NAFLD), effective diet and lifestyle treatments are imperative to curb this disease's impact. Our data suggests that insulin resistance is the strongest modifiable risk factor for having NAFLD. Additionally, genetic factors can interact with insulin resistance to multiplicatively increase risk of NAFLD. The investigators hypothesize that a very low-carbohydrate diet and behavioral support program may be able to achieve NAFLD reversal in adults with steatosis and/or mild fibrosis, especially in a subpopulation of rs738409-GG individuals. To prepare to test this, the investigators will conduct a pilot feasibility and acceptability trial of a 4-month online very low-carbohydrate, ketogenic (or keto) program in adults with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* have regular access to the internet
* MRI with liver steatosis but nor cirrhosis
* Able to consent and follow directions
* No physical limitations
* Physician approval to participate
* Able to attend in-person appointments in Ann Arbor
* Be identified based on information from the Michigan Genomics Initiative (MGI) database
* have elevated liver function tests

Exclusion Criteria:

* non-English speaking
* inability to complete baseline measurements
* a substance abuse, mental health, or medical condition that would interfere with participation (such as current chemotherapy, heart failure, kidney failure, Cushing's syndrome, etc.)
* pregnant or planning to get pregnant in the next 6 months
* type 1 diabetes
* non-NAFLD causes of elevated liver function tests
* planned or history of weight loss surgery
* vegan or vegetarian
* currently enrolled in a weight loss program or other investigative study that might conflict with this research
* taking medications known to cause weight gain or loss
* recent decompensation/hospitalization
* metal implants/inability to receive MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diet and Lifestyle Program
Started | 11
Completed | 9
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diet and Lifestyle Program
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.22 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Liver Fat Content Using Liver MRI-derived Proton Density Fat Fraction
Description: Measured with pre and post MRIs
Time Frame: 4 months
Population: We analyzed all participants with outcome data.
Measure: Mean (95% Confidence Interval); unit: percentage of liver lobe fat
Arm/Group | Diet and Lifestyle Program
Number analyzed (Participants) | 8
percentage of liver lobe fat | -7.06 [-15.5 to 1.37]

2. Secondary Outcome: Change in Liver Stiffness
Description: Change in liver stiffness as measured using Magnetic resonance (MR) elastography
Time Frame: 4 months
Population: We analyzed all participants with outcome data.
Measure: Mean (95% Confidence Interval); unit: kilopascals (kPa)
Arm/Group | Diet and Lifestyle Program
Number analyzed (Participants) | 6
kilopascals (kPa) | -0.33 [-0.82 to 0.17]

3. Secondary Outcome: Body Weight Change
Description: Measured with change in body weight
Time Frame: 4 months
Population: We analyzed all participants with outcome data.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Diet and Lifestyle Program
Number analyzed (Participants) | 9
kg | -10.69 [-13.37 to -8.00]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Diet and Lifestyle Program
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diet and Lifestyle Program (N=11)
diarrhea (Gastrointestinal disorders) | 1 (1)
flare up of dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
broken foot (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT05010070/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT05010070/ICF_000.pdf